CLINICAL TRIAL: NCT05393518
Title: Electroclinical Correlation of Anxiety, Evidences From Intracerebral Recordings
Brief Title: Electroclinical Correlation of Anxiety
Acronym: IRAnxNet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX 2020/63
Record Dates: First submitted 2022-03-29; First posted 2022-05-26 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Anxiety Disorder; Generalized Anxiety Disorder; Drug Resistant Epilepsy
Keywords: Focal epilepsy; Generalized Anxiety Disorder; Intracranial recordings; Stereoenectroencephalography; Coherence; Networks
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder; Drug Resistant Epilepsy; Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug resistant epilepsy with GAD (Experimental): Patients suffering from drug-resistant epilepsy and generalized anxiety disorders (GAD),explored by intracranial EEG (seteroelectroencephalography - SEEG) in Hospital
  Interventions: Behavioral: Anxiety-induced task; Behavioral: Neuropsychiatric assessment
- Drug resistant epilepsy without GAD (Active Comparator): Patients suffering from drug-resistant epilepsy without generalized anxiety disorders (GAD),explored by intracranial EEG (seteroelectroencephalography - SEEG) in Hospital
  Interventions: Behavioral: Anxiety-induced task; Behavioral: Neuropsychiatric assessment

INTERVENTIONS:
Behavioral: Anxiety-induced task — Subjects will be asked to describe their most anxious thoughts and write each of them in a detailed scenario. The scenarios will be based on the answers to the Worry and Anxiety Questionnaire, in order to validate the procedure by a standardized examination. During the task, the scenarios will be successively presented to the subjects, on a digital computer medium in written and oral format. Subjects will be asked to actively focus on these negative thoughts with maximum concern, without seeking to control their emotions.
Behavioral: Neuropsychiatric assessment — Screening for depression and anxiety

SUMMARY:
Anxiety disorders have the highest prevalence among mental disorders and cause considerable individual and financial costs. Current treatments do not relieve mental suffering of many patients. Understanding neurobiological mechanisms involved in pathological anxiety is a major scientific challenge.

DETAILED DESCRIPTION:
Functional imaging work has made it possible to identify the brain regions involved in anxiety disorders but is insufficient to study the pathophysiological mechanisms that cause anxiety symptoms. Brain regions involved in anxiety disorders are located deep in the human brain, and their electrophysiological study requires invasive recording methods.

Intracerebral electroencephalographic recordings (stereoelectroencephalography - sEEG) made for care in hospital before surgery in patients with drug-resistant epilepsy, offer this unique opportunity. Indeed, the brain regions involved in anxiety are among the structures registered to delimit the epilepticogenic zone, and 20% of patients with drug-resistant epilepsy suffer from an anxiety disorder.

This study propose to compare 15 patients suffering from drug-resistant epilepsy and generalized anxiety disorders (GAD), explored by intracranial sEEG, and 15 patients suffering from drug-resistant epilepsy without GAD ("controls"),explored by sEEG.

During sEEG patient will be proposed to undergo a custom-made behavioral task design to allow clinically-relevant anxiogenic exposure.

Patients will so be exposed to anxiety scenarios, while intracerebral sEEG, physiological stress parameters and the level of anxiety experienced will be monitored.

Electrophysiological parameters will be compared and correlated with clinical characteristics of the population and outcomes of the task.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Aged 18 to 65;
* With drug-resistant epilepsy
* Benefiting from a phase II pre-surgical assessment with intracerebral electrophysiological exploration by stereo-EEG
* Meeting the DSM-5 diagnostic criteria for generalized anxiety disorder ("pathological" population) or not meeting the DSM-5 diagnostic criteria for generalized anxiety disorder ("control" population)
* WAIS IV full scale IQ > 75 or IAG > 81
* Affiliate or beneficiary of a social security scheme
* Giving free, informed consent in writing and signed by the participant and the investigator

Exclusion Criteria:

* Being unable to give personal consent
* Be subject to a measure of legal protection (curatorship, guardianship) or placed under judicial protection;
* Suffer from a chronic delusional disorder (eg: schizophrenia);
* Have a moderate or high risk of suicide assessed using the corresponding section of the structured psychiatric interview called "Mini International Neuropsychiatric Interview" (M.I.N.I. 7.0) or a score > 2 on item 10 of the MADRS, assessing suicidal risk;
* Being pregnant or breastfeeding
* Have severe and / or decompensated somatic illness other than drug-resistant epilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2026-10-11 (Estimated); Study Completion 2026-10-11 (Estimated)

PRIMARY OUTCOMES:
Change in neuronal coherence in the frontolimbic network | Inclusion (Day 1)
  Change in neuronal coherence in the frontolimbic network between the basal condition and the expression of acute anxiety induced induced by exposure to an anxiety-inducing scenario between patients suffering from GAD and controls. Local brain activities tend to organize in oscillatory patterns. In order to determine if neurnal activities in frontal and limbic areas at similar oscillatory frequencies synchronize as a substrate or marker for anxiety, we will perform a coherence analysis. The coherence study estimates the consistency of the relative amplitude and phase of two signals in a given frequency spectrum, and will take its values in the interval [0.1]. The variation of coherence value will be compared between relevant epochs (anxiety-induced scenario and baseline) and between patients suffering from GAD and controls.

SECONDARY OUTCOMES:
Generalized Anxiety Disorders (GAD) severity score at The Penn State Worry Questionnaire (PSWQ) | Inclusion (Day 1)
  The Penn State Worry Questionnaire (PSWQ) is widely used in research and clinical practice to measure the tendency to worry in general. it includes 16 items assessing the general tendency to worry in adults. Patients are asked to respond spontaneously to 16 proposals by selecting the mention that best suits them
SEEG power spectrum changes | Inclusion (Day 1)
  the variation of power spectrum value or each frequency band (delta : [0.5 - 3] Hz, thêta : ]3 - 8] Hz, alpha : ]8 - 12] Hz, beta : ]12 - 25] Hz, gamma > 25 Hz) induced by exposure to an anxiety-inducing scenario will be compared between relevant epochs (anxiety-induced scenario and baseline) in patients suffering from GAD and controls, for each of the regions monitored.
Wechsler adult intelligent scale Score (WAIS-R full scale IQ) | Inclusion (Day 1)
  Test designed to measure the intellectual quotien (IQ) in terms of "verbal" and "performance". It is composed of 10 main mandatory subtests and 5 optional complementary subtests. These subtests are divided into four indices (verbal understanding, perceptual reasoning, working memory and processing speed). Scores ranged from 50 (minimum) to 150 (maximum).
Auditory and visual memory index (MEM IV) | Inclusion (Day 1)
  Normal values depend on its calibration according to the age of the subject and its level of education) is a test designed and validated to evaluate the learning and auditory and visual memory of a subject. They test different aspects of memory, including immediate recall, delayed recall, and recognition of visual and verbal stimuli.
Quality of life scale applied to epilepsy (QOLI-E 31) | Inclusion (Day 1)
  QOLI-E 31 containt 7 subtests evaluating the different health concepts (emotional well-being, social functioning, energy/fatigue, cognitive functioning, crisis anxiety, drug effects and overall quality of life).
Neurological Disorders Depression Inventoiry for Epilepsy (NDDI-E) | Inclusion (Day 1)
  Self-questionnaire of depressive disorder testing validated for epilepsy. Scores ranged from 0 (minimum) to 24(maximum). It consists of six items assessing depressive symptoms. Each item is rated on a 4-point Likert scale (1: never 2: rarely; 3: sometimes; 4: always or often, over the last two weeks). The total score is obtained by adding the score obtained for each item. A total score strictly higher than 15 must be suspected depressive syndrome. This questionnaire is also validated and has excellent psychometric properties (sensitivity and specificity) in the clinical population with epilepsy.
Generalized Anxiety Disorder 7- items (GAD-7) | Inclusion (Day 1)
  Self-test for anxiety disorders, including Generalized Anxiety Disorder. It consists of seven items assessing psychological and somatic anxiety symptoms. Each item is rated on a 4-point Likert scale (0: never; 1: several days; 2: more than half the time; 3: almost every day, over the last two weeks). The total score is obtained by adding the score obtained for each item (score ranging from 0 to 21). A total score strictly higher than 7 must make suspect a generalized anxiety disorder. If the score is higher than 7, it is advisable to have the diagnosis of TAG confirmed by a clinical psychiatric evaluation. This questionnaire is also validated and has excellent psychometric properties (sensitivity and specificity) in the clinical population with epilepsy.
Beck Depression Inventory (BDI) | Inclusion (Day 1)
  Scores ranged from 0 to 63. Self-assessment tool containing twenty-one elements that each describe one of the specific symptoms of depression. It can screen for recent depressive symptoms that have occurred in the past two weeks, and assess their severity. It can be used in subjects suffering from epilepsy. Each item is rated according to its intensity on a 4-point scale ranging from 0 (light intensity) to 3 (severe intensity). The maximum BDI score is 63 and the threshold for defining the presence of depression varies from 10 to 17, depending on the studies
Montgomery and Asberg Depression Rating Scale (MADRS) Score | Inclusion (Day 1)
  Hetero-questionnaire of mood assessment. It is rated by a trained clinician in its passing and consists of 10 items that each have a general definition and six degrees of severity of a symptom, with degrees 0, 2, 4 and 6 being themselves defined. The overall score (0 - 60) results from the addition of item scores.
State Anxiety Inventory (STAI) | Inclusion (Day 1)
  STAI is a two-part self-assessment questionnaire that independently assesses anxiety-trait and anxiety-state. They each include 20 items graduated in 4 degrees depending on their intensity or frequency. In the line-anxiety scale, the subject must indicate the point that best corresponds to the frequency of what he feels according to 4 degrees: 1 = almost never; 2 = sometimes; 3 = often; 4 = almost always. In the anxiety-state scale, the subject must indicate the point that best corresponds to the intensity of what he feels, also according to 4 degrees: 1 = no, 2 = rather no, 3 = rather yes, 4 = yes. The trait-anxiety scale is primarily used to assess the subject's usual anxiety temperament, while the state-anxiety scale is used to independently quantify current anxiety at the time of passing.
Beck Anxiety Inventory (BAI) | Inclusion (Day 1)
  utoquestionnaire that allows a quantitative estimate of the intensity of the anxiety feeling. It consists of 21 items of symptoms and attitudes resulting from panic and generalized anxiety disorders, evaluated over the last 7 days, graduated from 0 to 3 according to a Lickert scale
Hamilton Antiety rating Scale (HAM-A) Score | Inclusion (Day 1)
  Hetero-questionnaire intended to measure the severity of anxiety. It consists of 14 items corresponding to psychic and somatic anxiety symptoms noted on a 5-point Likert scale (0 - 4, in the increasing sense of severity). The overall score (0 - 56) results from the addition of the scores of items Hamilton et al. 1959. This is a classic trans-nosographic measure of the severity of anxiety. Its usefulness in this study consists of its evaluation by one. e clinician, while all other measures of anxiety are informed by patients
Analog Visual Scale (EVA) Anxiety score | Inclusion (Day 1)
  Anxiety self-assessessed during Anxiety task with Anxiety analog visual scale. (EVA-A)

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Aupy, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided